CLINICAL TRIAL: NCT00867048
Title: Strategic Timing of AntiRetroviral Treatment
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Copenhagen HIV Programme (CHIP) -- Copenhagen, Denmark (Unknown); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); ANRS, Emerging Infectious Diseases (Other Government); German Federal Ministry of Education and Research (Other Government); NEAT - European AIDS Treatment Network (Other); National Health and Medical Research Council, Australia (Other); National Institutes of Health Clinical Center (CC) (NIH); National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Abbott (Industry); Bristol-Myers Squibb (Industry); Gilead Sciences (Industry); GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry); Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0603M83587; U01AI068641 (NIH); 2008-006439-12 (EudraCT Number); NCT00821171 (obsolete NCT alias)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: HIV Infection
Keywords: highly active antiretroviral therapy (HAART); CD4 Count; Early Intervention; HIV; HIV Infection; HIV Infections; treatment naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early ART (Experimental): Initiate ART immediately following randomization
  Interventions: Drug: All licensed antiretroviral medications
- Deferred ART (Active Comparator): Defer ART until the CD4+ count declines to <350 cells/cu mm or AIDS develops
  Interventions: Drug: All licensed antiretroviral medications

INTERVENTIONS:
Drug: All licensed antiretroviral medications — In both arms, participants may be prescribed any licensed antiretroviral medication, in accordance with national treatment guidelines. The nature of the intervention is the timing of when to begin treatment with these medications, as described in the two treatment arms.

SUMMARY:
Objectives:

* To find out if the chance of developing a serious illness or of getting AIDS is less if patients start taking HIV medicines at a time when their cluster-of-differentiation-4 (CD4)+ cell count is still fairly high, instead of waiting until the CD4+ count is at the level where there is good evidence for starting medicines.
* To learn more about how a strategy of starting HIV medicines early might affect other aspects of care, such as the chances of developing other illnesses or resistance to HIV medicines, the frequency of doctor visits, the cost of medical care, and general health and satisfaction.

DETAILED DESCRIPTION:
Background:

* Most guidelines agree that if the number of your CD4+ cells (cells in your blood which help fight infection) drops below 350 cells/mm3, or if you have symptoms of AIDS, you should start taking HIV medicines. There are randomized trials that support this recommendation. (Randomized trials are usually considered the strongest form of evidence to support treatment decisions. Other studies, like observational studies, provide evidence too, but the evidence is often considered to be weaker than evidence from randomized trials. A randomized trial gives the most certain information about how well a treatment works because randomization makes sure each group is similar except for the treatment they receive.) Some experts believe that HIV treatment should be started even when the number of CD4+ cells is above 350 cells/mm3. For example, guidelines issued in the US in December 2009 include a new recommendation for starting HIV medicines if your CD4+ cell count is between 350 and 500 cells/mm3. However, this recommendation is based on information from observational studies, not randomized trials. We are doing this study to find out if the chances of getting a serious illness or of getting AIDS are less if people start taking HIV medicines at a time when their CD4+ cell counts are still fairly high, instead of waiting to take HIV medicines at a CD4+ count where there is good evidence for starting medicines.

Objectives:

* To find out if the chance of developing a serious illness or of getting AIDS is less if patients start taking HIV medicines at a time when their CD4+ cell count is still fairly high, instead of waiting until the CD4+ count is at the level where there is good evidence for starting medicines.
* To learn more about how a strategy of starting HIV medicines early might affect other aspects of care, such as the chances of developing other illnesses or resistance to HIV medicines, the frequency of doctor visits, the cost of medical care, and general health and satisfaction.

Eligibility:

* Patients 18 years of age and older who are infected with HIV, have CD4+ cell counts of greater than 500 cells/mm3, and who have never had antiretroviral therapy to treat HIV.

Design:

* Initial screening visits (2) to draw blood for CD4+ cell counts and provide a full medical history
* Patients will be randomly split into two groups:

Early: Patients will begin receiving HIV medications from the start of the study.

Deferred: Patients will begin to take HIV medications when the CD4 drops below 350 cells/mm3, or they develop AIDS or other symptoms of HIV infection.

* HIV medications for each patient will be determined by the study doctors.
* Evaluations during the treatment period:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Questions about daily life, including sexual behaviors.
* Blood and urine tests.
* Heart tests with electrocardiogram.
* Patients will return for evaluations at 1 and 4 months after randomization, and every 4 months thereafter for the duration of the study.

Substudies will take advantage of the START randomization to compare outcomes in people starting ART early vs. later.

The purpose of this randomized study is to determine whether immediate initiation of antiretroviral treatment (ART) is superior to deferral of ART until the CD4+ declines below 350 cells/mm(3) in terms of morbidity and mortality in HIV-1 (subsequently referred to as HIV) infected persons who are antiretroviral naive with a CD4+ count above 500 cells/mm(3).

The study will enroll an estimated 4,000 participants. Participants will be followed for at least 3 years after enrollment, to a common closing date.

Substudies will take advantage of the START randomization to compare outcomes in people starting ART early vs. later. These will measure outcomes that do not require the entire sample size of START to determine whether early ART is related to a difference in these outcomes over the course of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed informed consent
* HIV infection documented by a plasma HIV RNA viral load, rapid HIV test or any licensed* ELISA test; and confirmed by another test using a different method including but not limited to a rapid HIV test, Western Blot, HIV culture, HIV antigen, or HIV pro-viral DNA at any time prior to study entry.
* Age greater than or equal to 18 years
* Karnofsky performance score greater than or equal to 80 (an indication that the participant can perform normal activities)
* Perceived life expectancy of at least 6 months
* For women of child-bearing potential, willingness to use contraceptives as described in the product information of the ART drugs they are prescribed
* Two CD4+ cell counts greater than 500 cells/mm(3) at least 2 weeks apart within 60 days before randomization

  * The term licensed refers to an FDA-approved kit or, for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country. Confirmation of the initial test result must use a test method that is different than the one used for the initial assessment.

EXCLUSION CRITERIA:

* Any previous use of ART or interleukin-2 (IL-2)
* Diagnosis of any clinical AIDS event before randomization (including esophageal candidiasis and chronic Herpes simplex infection)
* Presence of HIV progression such as oral thrush, unexplained weight loss, or unexplained fever
* Cardiovascular event (myocardial infarction, angioplasty, coronary-artery bypass grafting, stroke) within 6 months before randomization
* Non-AIDS-defining cancer, excluding basal and squamous cell skin cancer, within 6 months before randomization
* Dialysis within 6 months before randomization
* Diagnosis of decompensated liver disease before randomization
* Current imprisonment, or compulsory detention (involuntary incarceration) for treatment of a psychiatric or physical illness
* Current pregnancy or breastfeeding (a negative serum or urine pregnancy test is required within 14 days before randomization for women of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4688 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Neaton, PhD, Principal Investigator — University of Minnesota; Abdel Babiker, PhD, Study Chair — Medical Research Council Clinical Trials Unit, London; Jens Lundgren, MD, DMSc, Study Chair — Copenhagen HIV Programme
Locations (218):
- United States (55):
  - University of Southern California, Alhambra, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - UCLA CARE-4-Families (LABAC CRS), Los Angeles, California
  - UCSD Mother-Child-Adolescent Program, San Diego, California
  - Naval Medical Center San Diego, San Diego, California
  - Denver Public Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Services Center, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Florida Department of Health in Orange County/Sunshine Care Center, Orlando, Florida
  - Infectious Diseases Associates NW FL, PA, Pensacola, Florida
  - Hillsborough County Health Deptment/University of South Florida, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Mt. Sinai Hospital, Chicago, Illinois
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Newland Immunology Center of Excellence (NICE), Southfield, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - New Jersey Medical School Adult Clinical Research Center, Newark, New Jersey
  - Cornell CRS, New York, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Regional Center for Infectious Disease, Greensboro, North Carolina
  - Wake County Human Services, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - The Research + Education Group - Portland, Portland, Oregon
  - The Research and Education Group at Portland VA Research Foundation, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Clinical Research Unit, Dallas, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston AIDS Research Team, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - San Antonio Military Health System, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - AIDS Resource Center of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - Hospital Nacional Profesor Alejandro Posadas, El Palomar, Buenos Aires
  - Hospital Interzonal General de Agudos Dr. Diego Paroissien, Isidro Casanova, Buenos Aires
  - CAICI (Instituto Centralizado de Assistencia e Investigacion Clinica Integral), Rosario, Santa Fe Province
  - FUNCEI, Buenos Aires
  - Fundacion IDEAA, Buenos Aires
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Rawson, Córdoba
  - CEIN, Neuquén
- Australia (13):
  - Burwood Road General Practice, Burwood, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sexual Health and HIV Service - Clinic 2, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
  - Centre Clinic, St Kilda, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Otto-Wagner-Spital SMZ /Baumgartner Hoehe, Vienna
  - University Vienna General Hospital, Vienna
- Belgium (4):
  - Institute of Tropical Medicine, Antwerp
  - Centre Hospitalier Universitaire St. Pierre (C.H.U. St. Pierre), Brussels
  - Universitaire Ziekenhuizen Gent, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
- Brazil (7):
  - Center for Infectious Diseases at the UFES, Vitória, Espírito Santo
  - SEI - Servi�os Especializados em Infectologia, Salvador, Estado de Bahia
  - Hospital Escola Sao Francisco de Assis - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Ipec/Fiocruz, Rio de Janeiro, Rio de Janeiro
  - Instituto de Infectologia Emilio Ribas - IIER, São Paulo, São Paulo
  - Centro de Referencia e Treinamento DST/Aids, São Paulo, São Paulo
  - Lim 56/Hcfmusp, São Paulo, São Paulo
- Fundacion Arriaran, Santiago, Chile
- Czechia (2):
  - University Hospital Plzen, CZ, Pilsen
  - Faculty Hospital Na Bulovce, Prague, Czech Rep., Prague
- Denmark (4):
  - Arhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet, Infektionsmedicinsk ambulatorium 8622, Copenhagen
  - Hvidovre University Hospital, Department of Infectious Diseases, Hvidovre
  - Odense University Hospital, Odense
- West Tallinn Central Hospital Infectious Diseases, Tallinn, Estonia
- Helsinki University Central Hospital, Div. of Infectious Diseases CRS, Helsinki, Finland
- France (12):
  - CHU de Besan�on - H�pital Jean-Minjoz, Besançon
  - CHU C�te de Nacre, Caen
  - H�pital Antoine Becl�re, Clamart
  - H�pital Henri Mondor, Créteil
  - H�pital de Bicetre, Le Kremlin-Bicêtre
  - Groupe Hospitalier Pitie-Salpetri�re, Paris
  - H�pital Europeen Georges Pompidou, Paris
  - H�pital H�tel Dieu, Paris
  - H�pital Saint-Antoine, Paris
  - H�pital Saint-Louis, Paris
  - H�pital Foch, Suresnes
  - Centre Hospitalier - H�pital Gustave Dron, Tourcoing
- Germany (17):
  - EPIMED-Gesellschaft fur epidemiologische und klinische Forschung in der MedizinmbH, Berlin
  - Gemeinschaftspraxis Jessen-Jessen-Stein, Berlin
  - Medizinische Universitatsklinik - Bonn, Immunologische Ambulanz CRS, Bonn
  - Klinik I fur Innere Medizin der Universitat zu Koln, Studienburo fur Infektiologie u. HIV, Cologne
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Erlangen, Erlangen
  - Klinik fur Dermatologie, Venerologie, Allergologie, Essen
  - Johann Wolfgang Goethe - University Hospital, Infektionsambulanz CRS, Frankfurt
  - ICH Study Center, Hamburg
  - Ifi - Studien und Projekte GmbH, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum der Universitat Munchen, Munich
  - Universitatsklinikum Regensburg, Regensburg
  - Universitatsklinikum Wurzburg, Medizinische Klinik und Poliklinik II, Schwerpunkt Infektiologie CRS, Würzburg
- Greece (6):
  - Attikon University General Hospital, Athens
  - Evangelismos General Hospital, Athens
  - Hippokration University General Hospital of Athens, Athens
  - Korgialenio-Benakio Hellenic Red Cross, Athens
  - Syngros Hospital, Athens
  - AHEPA University Hospital, Thessaloniki
- India (2):
  - Institute of Infectious Diseases, Pune, Maharashtra
  - YRGCARE Medical Centre VHS, Chennai CRS, Chennai, Tamil Nadu
- Mater Misericordiae University Hospital, Dublin, Ireland
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedale San Raffaele S.r.l., Milan, MI
  - Lazzaro Spallanzani IRCSS, Rome, RM
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia
- Serefo/Cesac Mali, Bamako, Mali
- INCMNSZ (Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran), Tlalpan, Mexico
- University Hospital Centre Ibn Rochd, Casablanca, Morocco
- Institute of Human Virology-Nigeria (IHVN), Abuja, Federal Capital Territory, Nigeria
- Oslo University Hospital, Ulleval, Oslo, Norway
- Peru (5):
  - Via Libre, Lima
  - Asociacion Civil IMPACTA Salud y Educacion, Lima
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
  - Asociacion Civil Impacta Salud y Educacion - Sede San Miguel, Lima
- Poland (3):
  - Uniwersytecki Szpital Kliniczny, Bialystok
  - Wojewodzki Szpital Zakazny, Warsaw
  - EMC Instytut Medyczny SA, Wroclaw
- Portugal (4):
  - Hospital Curry Cabral, Lisbon
  - Hospital de Egas Moniz, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Joaquim Urbano, Porto
- Puerto Rico (3):
  - San Juan Hospital, Rio Piedras
  - University of Puerto Rico Pediatric Research Site, San Juan
  - Puerto Rico-AIDS Clinical Trials Unit (PR-ACTU), San Juan
- South Africa (5):
  - Desmond Tutu HIV Foundation Clinical Trials Unit, Cape Town
  - Durban International Clinical Research Site (WWH), Durban
  - Durban International Clinical Research Site, Durban
  - CHRU, Johannesburg
  - 1 Military Hospital, Pretoria
- Spain (12):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital La Princesa, Internal Medicine and Infectious Disease Service CRS, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitari Mutua Terrassa, Terrassa
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Complejo Hospitalario Xeral Cies, Vigo
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Malmo
- Switzerland (4):
  - University Hospital Basel, Basel
  - Bern University Hospital, Bern
  - Unite VIH/SIDA Geneva, Geneva
  - University Hospital Zurich, Zurich
- Thailand (9):
  - Chulalongkorn University Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok Noi
  - Sanpatong Hospital, Chiang Mai
  - Research Institute for Health Sciences (RIHES), Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Chonburi Regional Hospital, Chon Buri
  - Khon Kaen University, Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi
- Uganda (2):
  - MRC/UVRI Research Unit on AIDS, Entebbe
  - Joint Clinical Research Center (JCRC), Kampala
- United Kingdom (21):
  - Royal Berkshire Hospital, Reading, Berkshire
  - The James Cook University Hospital, Middlesbrough, Cleveland
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Belfast Health and Social Care Trust (RVH), Belfast, Northern Ireland
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Coventry and Warwickshire NHS partnership Trust, Coventry, West Midlands
  - Southmead Hospital, Bristol
  - Gloucestershire Royal Hospital, Gloucester
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St.Thomas' NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - Chelsea and Westminster Hospital, London
  - St. George's Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - University College London Medical School, London
  - North Manchester General Hospital, Manchester

REFERENCES:
- [Background] Babiker AG, Emery S, Fatkenheuer G, Gordin FM, Grund B, Lundgren JD, Neaton JD, Pett SL, Phillips A, Touloumi G, Vjechaj MJ; INSIGHT START Study Group. Considerations in the rationale, design and methods of the Strategic Timing of AntiRetroviral Treatment (START) study. Clin Trials. 2013;10(1 Suppl):S5-S36. doi: 10.1177/1740774512440342. Epub 2012 Apr 30. PMID 22547421
- [Result] INSIGHT START Study Group; Lundgren JD, Babiker AG, Gordin F, Emery S, Grund B, Sharma S, Avihingsanon A, Cooper DA, Fatkenheuer G, Llibre JM, Molina JM, Munderi P, Schechter M, Wood R, Klingman KL, Collins S, Lane HC, Phillips AN, Neaton JD. Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection. N Engl J Med. 2015 Aug 27;373(9):795-807. doi: 10.1056/NEJMoa1506816. Epub 2015 Jul 20. PMID 26192873
- [Derived] MacDonald DM, Samorodnitsky S, Wendt CH, Baker JV, Collins G, Kruk M, Lock EF, Paredes R, Poongulali S, Weise DO, Winston A, Wood R, Kunisaki KM; INSIGHT START Pulmonary Substudy Group. Pneumoproteins and biomarkers of inflammation and coagulation do not predict rapid lung function decline in people living with HIV. Sci Rep. 2023 Mar 23;13(1):4749. doi: 10.1038/s41598-023-29739-x. PMID 36959289
- [Derived] Gabrielaite M, Bennedbaek M, Rasmussen MS, Kan V, Furrer H, Flisiak R, Losso M, Lundgren JD; INSIGHT START Study Group; Marvig RL. Deep-sequencing of viral genomes from a large and diverse cohort of treatment-naive HIV-infected persons shows associations between intrahost genetic diversity and viral load. PLoS Comput Biol. 2023 Jan 3;19(1):e1010756. doi: 10.1371/journal.pcbi.1010756. eCollection 2023 Jan. PMID 36595537
- [Derived] Gabrielaite M, Bennedbaek M, Zucco AG, Ekenberg C, Murray DD, Kan VL, Touloumi G, Vandekerckhove L, Turner D, Neaton J, Lane HC, Safo S, Arenas-Pinto A, Polizzotto MN, Gunthard HF, Lundgren JD, Marvig RL. Human Immunotypes Impose Selection on Viral Genotypes Through Viral Epitope Specificity. J Infect Dis. 2021 Dec 15;224(12):2053-2063. doi: 10.1093/infdis/jiab253. PMID 33974707
- [Derived] Ghazi L, Baker JV, Sharma S, Jain MK, Palfreeman A, Necsoi C, Murray DD, Neaton JD, Drawz PE. Role of Inflammatory Biomarkers in the Prevalence and Incidence of Hypertension Among HIV-Positive Participants in the START Trial. Am J Hypertens. 2020 Jan 1;33(1):43-52. doi: 10.1093/ajh/hpz132. PMID 31800000
- [Derived] Lampe FC, Rodger AJ, Burman W, Grulich A, Friedland G, Sadr WE, Neaton J, Corbelli GM, Emery S, Molina JM, Orkin C, Gatell J, Gerstoft J, Ruxrungtham K, Barbosa de Souza M, Phillips AN; INSIGHT START Study Group. Impact of early antiretroviral treatment on sexual behaviour: a randomised comparison. AIDS. 2019 Dec 1;33(15):2337-2350. doi: 10.1097/QAD.0000000000002359. PMID 31764099
- [Derived] Wyman Engen N, Huppler Hullsiek K, Belloso WH, Finley E, Hudson F, Denning E, Carey C, Pearson M, Kagan J. A randomized evaluation of on-site monitoring nested in a multinational randomized trial. Clin Trials. 2020 Feb;17(1):3-14. doi: 10.1177/1740774519881616. Epub 2019 Oct 24. PMID 31647325
- [Derived] Castillo-Mancilla JR, Phillips AN, Neaton JD, Neuhaus J, Sharma S, Baker JV, Collins S, Mannheimer S, Pett S, Touzeau-Romer V, Polizzotto MN, Lundgren JD, Gardner EM; INSIGHT START Study Group. Incomplete ART adherence is associated with higher inflammation in individuals who achieved virologic suppression in the START study. J Int AIDS Soc. 2019 Jun;22(6):e25297. doi: 10.1002/jia2.25297. PMID 31250552
- [Derived] Borges AH, Neuhaus J, Sharma S, Neaton JD, Henry K, Anagnostou O, Staub T, Emery S, Lundgren JD; INSIGHT SMART; START Study Groups. The Effect of Interrupted/Deferred Antiretroviral Therapy on Disease Risk: A SMART and START Combined Analysis. J Infect Dis. 2019 Jan 7;219(2):254-263. doi: 10.1093/infdis/jiy442. PMID 30032171
- [Derived] Molina JM, Grund B, Gordin F, Williams I, Schechter M, Losso M, Law M, Ekong E, Mwelase N, Skoutelis A, Wiselka MJ, Vandekerckhove L, Benfield T, Munroe D, Lundgren JD, Neaton JD; INSIGHT START study group. Which HIV-infected adults with high CD4 T-cell counts benefit most from immediate initiation of antiretroviral therapy? A post-hoc subgroup analysis of the START trial. Lancet HIV. 2018 Apr;5(4):e172-e180. doi: 10.1016/S2352-3018(18)30003-1. Epub 2018 Jan 16. PMID 29352723
- [Derived] Ronit A, Sharma S, Baker JV, Mngqibisa R, Delory T, Caldeira L, Ndembi N, Lundgren JD, Phillips AN; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) Strategic Timing of Antiretroviral Treatment (START) Study Group. Serum Albumin as a Prognostic Marker for Serious Non-AIDS Endpoints in the Strategic Timing of Antiretroviral Treatment (START) Study. J Infect Dis. 2018 Jan 17;217(3):405-412. doi: 10.1093/infdis/jix350. PMID 29244111
- [Derived] Baker JV, Sharma S, Achhra AC, Bernardino JI, Bogner JR, Duprez D, Emery S, Gazzard B, Gordin J, Grandits G, Phillips AN, Schwarze S, Soliman EZ, Spector SA, Tambussi G, Lundgren J; INSIGHT (International Network for Strategic Initiatives in Global HIV Trials) START (Strategic Timing of Antiretroviral Treatment) Study Group. Changes in Cardiovascular Disease Risk Factors With Immediate Versus Deferred Antiretroviral Therapy Initiation Among HIV-Positive Participants in the START (Strategic Timing of Antiretroviral Treatment) Trial. J Am Heart Assoc. 2017 May 22;6(5):e004987. doi: 10.1161/JAHA.116.004987. PMID 28533305
- [Derived] Grady C, Touloumi G, Walker AS, Smolskis M, Sharma S, Babiker AG, Pantazis N, Tavel J, Florence E, Sanchez A, Hudson F, Papadopoulos A, Emanuel E, Clewett M, Munroe D, Denning E; INSIGHT START Informed Consent Substudy Group. A randomized trial comparing concise and standard consent forms in the START trial. PLoS One. 2017 Apr 26;12(4):e0172607. doi: 10.1371/journal.pone.0172607. eCollection 2017. PMID 28445471
- [Derived] O'Connor J, Vjecha MJ, Phillips AN, Angus B, Cooper D, Grinsztejn B, Lopardo G, Das S, Wood R, Wilkin A, Klinker H, Kantipong P, Klingman KL, Jilich D, Herieka E, Denning E, Abubakar I, Gordin F, Lundgren JD; INSIGHT START study group. Effect of immediate initiation of antiretroviral therapy on risk of severe bacterial infections in HIV-positive people with CD4 cell counts of more than 500 cells per muL: secondary outcome results from a randomised controlled trial. Lancet HIV. 2017 Mar;4(3):e105-e112. doi: 10.1016/S2352-3018(16)30216-8. Epub 2017 Jan 5. PMID 28063815
- [Derived] Larson GS, Carey C, Grarup J, Hudson F, Sachi K, Vjecha MJ, Gordin F; INSIGHT Group. Lessons learned: Infrastructure development and financial management for large, publicly funded, international trials. Clin Trials. 2016 Apr;13(2):127-36. doi: 10.1177/1740774515625974. Epub 2016 Feb 8. PMID 26908541
- [Derived] Carr A, Grund B, Neuhaus J, Schwartz A, Bernardino JI, White D, Badel-Faesen S, Avihingsanon A, Ensrud K, Hoy J; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Prevalence of and risk factors for low bone mineral density in untreated HIV infection: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):137-46. doi: 10.1111/hiv.12242. PMID 25711332
- [Derived] Matthews GV, Neuhaus J, Bhagani S, Mehta SH, Vlahakis E, Doroana M, Naggie S, Arenas-Pinto A, Peters L, Rockstroh JK; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Baseline prevalence and predictors of liver fibrosis among HIV-positive individuals: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(Suppl 1):129-36. doi: 10.1111/hiv.12241. PMID 25711331
- [Derived] Kunisaki KM, Niewoehner DE, Collins G, Nixon DE, Tedaldi E, Akolo C, Kityo C, Klinker H, La Rosa A, Connett JE; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Pulmonary function in an international sample of HIV-positive, treatment-naive adults with CD4 counts > 500 cells/muL: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 0):119-28. doi: 10.1111/hiv.12240. PMID 25711330
- [Derived] Baker JV, Engen NW, Huppler Hullsiek K, Stephan C, Jain MK, Munderi P, Pett S, Duprez D; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Assessment of arterial elasticity among HIV-positive participants with high CD4 cell counts: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):109-18. doi: 10.1111/hiv.12239. PMID 25711329
- [Derived] Wright EJ, Grund B, Cysique LA, Robertson KR, Brew BJ, Collins G, Shlay JC, Winston A, Read TR, Price RW; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Factors associated with neurocognitive test performance at baseline: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1:97-108. doi: 10.1111/hiv.12238. PMID 25711328
- [Derived] Lifson AR, Grandits GA, Gardner EM, Wolff MJ, Pulik P, Williams I, Burman WJ; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Quality of life assessment among HIV-positive persons entering the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):88-96. doi: 10.1111/hiv.12237. PMID 25711327
- [Derived] Baxter JD, Dunn D, White E, Sharma S, Geretti AM, Kozal MJ, Johnson MA, Jacoby S, Llibre JM, Lundgren J; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Global HIV-1 transmitted drug resistance in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):77-87. doi: 10.1111/hiv.12236. PMID 25711326
- [Derived] Rodger AJ, Lampe FC, Grulich AE, Fisher M, Friedland G, Phanuphak N, Bogner JR, Pereira LC, Rietmeijer C, Burman W, Phillips AN; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Transmission risk behaviour at enrolment in participants in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 0):64-76. doi: 10.1111/hiv.12235. PMID 25711325
- [Derived] Achhra AC, Mocroft A, Ross MJ, Ryom L, Lucas GM, Furrer H, Neuhaus J, Somboonwit C, Kelly M, Gatell JM, Wyatt CM; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Kidney disease in antiretroviral-naive HIV-positive adults with high CD4 counts: prevalence and predictors of kidney disease at enrolment in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):55-63. doi: 10.1111/hiv.12234. PMID 25711324
- [Derived] Soliman EZ, Sharma S, Arasteh K, Wohl D, Achhra A, Tambussi G, O'Connor J, Stein JH, Duprez DA, Neaton JD, Phillips A; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Baseline cardiovascular risk in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 0):46-54. doi: 10.1111/hiv.12233. PMID 25711323
- [Derived] Law MG, Achhra A, Deeks SG, Gazzard B, Migueles SA, Novak RM, Ristola M; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Clinical and demographic factors associated with low viral load in early untreated HIV infection in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):37-45. doi: 10.1111/hiv.12232. PMID 25711322
- [Derived] Sharma S, Babiker AG, Emery S, Gordin FM, Lundgren JD, Neaton JN, Bakowska E, Schechter M, Wiselka MJ, Wolff MJ; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Demographic and HIV-specific characteristics of participants enrolled in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):30-6. doi: 10.1111/hiv.12231. PMID 25711321
- [Derived] Denning E, Sharma S, Smolskis M, Touloumi G, Walker S, Babiker A, Clewett M, Emanuel E, Florence E, Papadopoulos A, Sanchez A, Tavel J, Grady C; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Reported consent processes and demographics: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):24-9. doi: 10.1111/hiv.12230. PMID 25711320
- [Derived] Grarup J, Rappoport C, Engen NW, Carey C, Hudson F, Denning E, Sharma S, Florence E, Vjecha MJ; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Challenges, successes and patterns of enrolment in the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(Suppl Suppl 1):14-23. doi: 10.1111/hiv.12229. PMID 25711319
- [Derived] Geffen N, Aagaard P, Corbelli GM, Meulbroek M, Peavy D, Rappoport C, Schwarze S, Collins S; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) Community Advisory Board. Community perspective on the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):10-3. doi: 10.1111/hiv.12228. PMID 25711318
- [Derived] INSIGHT Strategic Timing of AntiRetroviral Treatment (START) Study Group; Lundgren J, Babiker A, Gordin F, Emery S, Fatkenheuer G, Molina JM, Wood R, Neaton JD. Why START? Reflections that led to the conduct of this large long-term strategic HIV trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):1-9. doi: 10.1111/hiv.12227. No abstract available. PMID 25711317
- [Derived] Kunisaki KM, Quick H, Baker JV. HIV antiretroviral therapy reduces circulating surfactant protein-D levels. HIV Med. 2011 Oct;12(9):580-1. doi: 10.1111/j.1468-1293.2011.00920.x. No abstract available. PMID 21951596
- See also: INSIGHT network website, including information on the START trial — http://www.insight-trials.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Early ART: Initiate ART immediately following randomization
  All licensed antiretroviral medications: In both arms, participants may be prescribed any licensed antiretroviral medication, in accordance with national treatment guidelines. The nature of the intervention is the timing of when to begin treatment with these medications, as described in the two treatment arms.
  ART dosage and frequency were based on clinical decision in accordance with local/national prescribing guidelines.
- Deferred ART: Defer ART until the CD4+ count declines to <350 cells/cu mm or AIDS develops
  All licensed antiretroviral medications: In both arms, participants may be prescribed any licensed antiretroviral medication, in accordance with national treatment guidelines. The nature of the intervention is the timing of when to begin treatment with these medications, as described in the two treatment arms.
  ART dosage and frequency were based on clinical decision in accordance with local/national prescribing guidelines.
Period: Overall Study
Arm/Group | Early ART | Deferred ART
Started | 2326 | 2362
Completed | 2325 | 2359
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early ART | Deferred ART | Total
Number analyzed (Participants) | 2326 | 2362 | 4688
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2308 | 2345 | 4653
  >=65 years | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.2) | 36.8 (10.1) | 36.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 624 | 635 | 1259
  Male | 1702 | 1727 | 3429
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 197 | 190 | 387
  Native Hawaiian or Other Pacific Islander | 701 | 704 | 1405
  Black or African American | 1025 | 1084 | 2109
  White | 3 | 6 | 9
  More than one race | 308 | 303 | 611
  Unknown or Not Reported | 91 | 74 | 165

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of AIDS, Serious Non-AIDS Diagnoses, and All-cause Mortality
Time Frame: full follow-up, 9.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 2325 | 2359
Participants | 133 | 215

2. Secondary Outcome: AIDs or AIDs Related Death
Description: participant count
Time Frame: full follow-up, 9.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 2325 | 2359
Participants | 31 | 83

3. Secondary Outcome: Specific Non-AIDS Diagnoses
Time Frame: full follow-up, 9.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 2325 | 2359
Participants | 107 | 137

4. Secondary Outcome: Death, All-cause Mortality
Description: Count of participants
Time Frame: full follow-up, 9.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 2325 | 2359
Participants | 66 | 85

5. Secondary Outcome: Quality of Life- Mean Change From Baseline in a Visual Analog Scale (VAS) for Perceived Current Health
Description: Mean change from baseline of the VAS. This was a single data item where participants self-reported their perceived current state of health on a scale of 0-100 (0=worst possible and 100=best possible).
Time Frame: 4.5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 2253 | 2287
units on a scale | 1.8 (8.6) | 0.22 (8.7)

6. Secondary Outcome: Transmission Risk Behavior Outcome 1
Description: Proportion of participants identifying as men who have sex with men (MSM) engaging in condomless sex with HIV serodifferent partners (CLS-D) at study month 12. Participant completed a self-reported questionnaire on transmission risk behavior during the "past two months" at the month 12 visit following randomization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 1236 | 1187
Participants | 156 | 155

7. Secondary Outcome: Change in Neurocognitive Function (in a Subset of Participants)
Description: Mean change from baseline of the QNPZ-8 score. In the Neurology substudy of START, participants were administered a neuropsychological test battery of 8 tests (grooved peg board, finger tapping, Color Trails 1 and 2, Semantic Verbal Fluency, WAIS III Digit Symbol, HVLT-R Learning, HVLT-R Delayed Recall). Test scores were standardized to z-scores using baseline values as reference such that baseline values had a mean of 0 and standard deviation of 1. Test scores were standardized to z-scores using baseline values as reference such that baseline values had a mean of 0 and standard deviation of 1. Z-scores > 0 indicate improvement over baseline levels. The quantitative neuropsychological performance z-score (QNPZ-8) was the mean of the z-scores across the the 8 tests. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 291 | 301
units on a scale | 0.19 [0.16 to 0.23] | 0.21 [0.18 to 0.25]

8. Secondary Outcome: Large Artery Elasticity (in a Subset of Participants)
Description: Mean change from baseline in large arterial elasticity. In the Arterial Elasticity substudy of START, participants had non-invasive measurements of radial artery blood pressure waveforms recorded at baseline, study months 4, 8, and 12, and then annually. Small arterial elasticity (SAE) and large arterial elasticity (LAE) were derived from analysis of the diastolic pulse waveform. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (Full Range); unit: mL/mmHg x 10
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 178 | 154
mL/mmHg x 10 | 0.27 [0.02 to 0.53] | 0.8 [0.52 to 1.07]

9. Secondary Outcome: Rate of Lung Function Decline (in a Subset of Participants) Among
Description: Rate of lung function decline (slope of forced expiratory volume (FEV1)) over follow-up among self-reported smokers at study entry. In the pulmonary substudy of START, participants had post-bronchodilator spirometry measures collected at baseline and annually. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (95% Confidence Interval); unit: mL/yr
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 135 | 156
mL/yr | -36.6 [-51 to -22.3] | -38.8 [-52.8 to -24.8]

10. Secondary Outcome: Changes in Bone Mineral Density (in a Subset of Participants) Measure 1
Description: Mean percent change from baseline in bone mineral density at the spine. In the bone mineral density (BMD) substudy of START, participants underwent dual-enery x-ray absorptionmetry (DXA) to measure BMD at the spine and hip at baseline and annually. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 201 | 210
percent | -1.8 [-2.3 to -1.4] | -0.9 [-1.3 to -0.4]

11. Secondary Outcome: Transmission Risk Behavior Outcome 2
Description: Percentage of participants identifying as hetrosexual engaging in condomless sex with HIV serodifferent partners (CLS-D) at study month 12. Participant completed a self-reported questionnaire on transmission risk behavior during the "past two months" at the month 12 visit following randomization.
Time Frame: 12 month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 934 | 964
Participants | 101 | 80

12. Secondary Outcome: Small Artery Elasticity (in a Subset of Participants)
Description: Mean change from baseline in small arterial elasticity. In the Arterial Elasticity substudy of START, participants had non-invasive measurements of radial artery blood pressure waveforms recorded at baseline, study months 4, 8, and 12, and then annually. Small arterial elasticity (SAE) and large arterial elasticity (LAE) were derived from analysis of the diastolic pulse waveform. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (Full Range); unit: mL/mmHg x 10
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 178 | 154
mL/mmHg x 10 | -0.23 [-0.41 to -0.06] | -0.18 [-0.37 to 0.01]

13. Secondary Outcome: Rate of Lung Function Decline (in a Subset of Participants) Among Non-smokers
Description: Rate of lung function decline (slope of forced expiratory volume (FEV1)) over follow-up among self-reported non-smokers at study entry. In the pulmonary substudy of START, participants had post-bronchodilator spirometry measures collected at baseline and annually. Analyses were by intention-to-treat principles.
Time Frame: 4.5 years
Measure: Mean (95% Confidence Interval); unit: mL/yr
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 383 | 353
mL/yr | -26.9 [-34.1 to -19.8] | -22.8 [-30.4 to -15.3]

14. Secondary Outcome: Changes in Bone Mineral Density (in a Subset of Participants) Measure 2
Description: as for outcome 10
Time Frame: 4.5 years
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Early ART | Deferred ART
Number analyzed (Participants) | 200 | 210
percent | -2.8 [-3.3 to -2.2] | -1.7 [-2.2 to -1.1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality assessed up to a median of 9.3 years. Serious Adverse Events were assessed for a median of 5.5 years
Description: Non-serious adverse events were not collected. Of the total number of participants randomized, 4 participants were found out to be HIV negative. Those participants were all administratively withdrawn from the study and were not followed for adverse events. Adverse events reported are those collected as "Serious Events" which were only collected through 31 December 2017. Deaths were collected through full follow-up and are reported separately under Outcome 4.
Arm/Group | Early ART | Deferred ART
All-Cause Mortality (participants affected / at risk) | 66/2325 | 85/2359
Serious Adverse Events (participants affected / at risk) | 428/2325 | 500/2359
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early ART (N=2325) | Deferred ART (N=2359)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 7 (7)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 8 (8) | 6 (6)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (6) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (3) | 1 (1)
Foetal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Subvalvular aortic stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Alagille syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anencephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Disorder of orbit (Eye disorders) | 1 (1) | 0 (0)
Opsoclonus myoclonus (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (5) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 4 (6)
Proctitis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (5)
Chills (General disorders) | 1 (1) | 0 (0)
Complication of device insertion (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 12 (12)
Drowning (General disorders) | 0 (0) | 2 (2)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Impaired self-care (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Necrobiosis (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (3) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 11 (12)
Strangulated hernia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 5 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholelithiasis migration (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 3 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (4) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 7 (7) | 4 (4)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Acute hepatitis C (Infections and infestations) | 4 (4) | 2 (2)
Anal abscess (Infections and infestations) | 5 (6) | 13 (14)
Appendicitis (Infections and infestations) | 24 (24) | 17 (17)
Appendicitis perforated (Infections and infestations) | 1 (3) | 0 (0)
Arteriovenous graft site abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (2) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 1 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Campylobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 5 (5) | 10 (12)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (4)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Embolic pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 4 (4) | 1 (1)
Epiglottic abscess (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 4 (4)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 3 (3)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 10 (10)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 2 (3) | 1 (1)
HIV associated nephropathy (Infections and infestations) | 0 (0) | 1 (1)
HIV peripheral neuropathy (Infections and infestations) | 0 (0) | 1 (2)
Hepatitis A (Infections and infestations) | 6 (6) | 4 (4)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex necrotising retinopathy (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 7 (7)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Lymph node abscess (Infections and infestations) | 0 (0) | 1 (1)
Lymphogranuloma venereum (Infections and infestations) | 1 (1) | 1 (1)
Malaria (Infections and infestations) | 4 (4) | 9 (10)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 2 (2)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Mononucleosis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium abscessus infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 2 (2) | 6 (7)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 2 (2) | 4 (4)
Osteomyelitis (Infections and infestations) | 1 (3) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Parotid abscess (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 2 (2) | 4 (6)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 3 (3) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 2 (2) | 1 (1)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 0 (0)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 2 (2)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Rubella (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 6 (6)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 3 (3)
Shigella infection (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Strongyloidiasis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 3 (3)
Syphilis (Infections and infestations) | 0 (0) | 4 (4)
Tertiary syphilis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 3 (3)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (7) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (5)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture of penis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Testicular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (12)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extragonadal primary seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Testicular germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 5 (6)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Drug withdrawal convulsions (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 3 (3) | 2 (2)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 2 (2)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Postictal state (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 3 (3)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (5) | 2 (2)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 2 (2)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (2)
Alcoholism (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (5)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 3 (3) | 1 (1)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 1 (2)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 5 (5)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 8 (9) | 13 (18)
Depression suicidal (Psychiatric disorders) | 3 (3) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 2 (2)
Major depression (Psychiatric disorders) | 7 (8) | 3 (3)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (3) | 2 (3)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 2 (3)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 3 (3)
Substance-induced mood disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 3 (6) | 3 (4)
Suicidal ideation (Psychiatric disorders) | 14 (22) | 16 (22)
Suicide attempt (Psychiatric disorders) | 24 (34) | 20 (22)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 6 (6)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 3 (3)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 4 (4)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (8)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Xanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Homicide (Social circumstances) | 1 (1) | 0 (0)
Substance use (Social circumstances) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortitis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 3 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT00867048/Prot_SAP_ICF_000.pdf